CLINICAL TRIAL: NCT06932471
Title: A Multicenter, Single-arm, Open-label Phase III Study to Evaluate Efficacy and Safety of MY008211A Tablets in Patients With PNH and Residual Anemia, Despite Treatment With Anti-C5 Antibody.
Brief Title: Study of Safety and Efficacy of MY008211A in Patients With Residual Anemia Despite Anti-C5 Antibody Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MY008211A-PNH-3-01
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MY008211A tablets (Experimental): MY008211A tablets 400mg BID
  Interventions: Drug: MY008211A tablets

INTERVENTIONS:
Drug: MY008211A tablets — MY008211A tablets Participants will receive MY008211A at a dose of 400 mg orally b.i.d
  Other Names: MY008211A

SUMMARY:
The main purpose of this study is to evaluate the efficacy of MY008211A in PNH patients with residual anemia despite treatment with anti-C5 antibody.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label phase III clinical trial. The purpose of this study is to determine whether MY008211A is efficacious and safe for the treatment of PNH patients Who Are Still Anemia After Anti-C5 Antibody Treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age and BMI ≥ 18.0 kg/m2 with a diagnosis of PNH confirmed by high-sensitivity flow cytometry with clone size ≥ 10%.
2. Stable regimen of anti-C5 antibody treatment for at least 6 months before treatment, and Hb was still < 100 g/L.
3. The average hemoglobin level of at least two tests in 4 months before screening < 100 g/L.
4. The average hemoglobin level of two tests in the central laboratory during screening < 100 g/L.
5. Vaccination against Neisseria meningitidis infection is required prior to the start of study treatment. If not received previously, vaccination against Streptococcus pneumoniae and Haemophilus influenzae infections should be given.

Exclusion Criteria:

1. Patients with reticulocytes <100x10^9/L; platelets <30x10^9/L; neutrophils <0.5x10^9/L.
2. History of recurrent invasive infections caused by encapsulated organisms,e.g. meningococcus or pneumococcus.
3. Known or suspected hereditary complement deficiency.
4. Previous bone marrow or hematopoietic stem cell transplantation.
5. Previous splenectomy.
6. A history of malignancy within 5 years before screening, except cured local basal cell carcinoma of the skin and carcinoma in situ of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of Participants With Sustained Hemoglobin Levels of ≥ 120 g/L in the Absence of Red Blood Cell Transfusions (defined as no red blood cell infusion after D14 to D168) | between Day 126 and Day 168
  The proportion of patients with sustained hemoglobin levels ≥ 120 g/L among those without RBC transfusion.

SECONDARY OUTCOMES:
The proportion of subjects with an increase in hemoglobin concentration ≥ 20 g/L from baseline among subjects who do not receive RBC transfusion (defined as no red blood cell infusion after D14 to D168) | between Day 126 and Day 168
  Proportion of participants achieving a sustained increase from baseline in hemoglobin levels of ≥ 20 g/L assessed among those without RBC transfusion.
Change From Baseline in Hemoglobin | between Day 126 and Day 168
  Change in hemoglobin concentration from baseline in patients without RBC transfusion.
The proportion of patients with LDH < 1.5 ULN among those without RBC transfusion. | between Day 126 and Day 168
  The proportion of patients with hemolysis controlled (defined as LDH < 1.5 ULN) among those without RBC transfusion.
Change (Expressed as Percentages) in LDH level from baseline | between Day 126 and Day 168
  Change (Expressed as Percentages) in LDH level from baseline
Change in reticulocyte count from baseline | between Day 126 and Day 168
  Change in reticulocyte count from baseline
The proportion of patients without RBC transfusion | between Day 14 and Day 168
  The proportion of patients without RBC transfusion.
Change in FACIT-F score from baseline | between Day 126 and Day 168
  Change in FACIT-Fatigue score from baseline. The FACIT-Fatigue is a 13-item questionnaire with support for its validity and reliability in PNH that assesses patient self-reported fatigue and its impact on daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F Scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
The Clinical BTH Rate | between Day 1 and Day 168
  The Clinical BTH Rate
The Major Adverse Vascular Events Rate | between Day 1 and Day 168
  The Major Adverse Vascular Events Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital (PUMCH)., Beijing, Beijing Municipality, China